CLINICAL TRIAL: NCT03636984
Title: Efficacy and Safety Study of Anbainuo in Chinese Patients With Rheumatoid Arthritis/ Ankylosing Spondylitis in the Real World: a Prospective, Open-label, Multi-center Observational Study
Brief Title: Efficacy and Safety Study of Anbainuo in Chinese Patients With RA/AS in the Real World
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Bioinno-ABN-2018001
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing | interventions — Anbainuo protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rheumatoid arthritis patients: subjects with rheumatoid arthritis would be administered with recombinant TNF-α receptor: IgG Fc fusion protein （Anbainuo）50 mg peer week for 3 to 6 months until reaching clinical remission or low disease activity. Then the application of Anbainuo would be continued for 6 months. If the subjects did not reach clinical remission or low disease activity in 6 months, the treatment should be considered as invalid.
  Interventions: Drug: recombinant TNF-α receptor: IgG Fc fusion protein
- ankylosing spondylitis patients: subjects with ankylosing spondylitis would be administered with recombinant TNF-α receptor: IgG Fc fusion protein （Anbainuo）50 mg peer week for 3 to 6 months until reaching clinical remission or low disease activity. Then the application of Anbainuo would be continued for 6 months. If the subjects did not reach clinical remission or low disease activity in 6 months, the treatment should be considered as invalid.
  Interventions: Drug: recombinant TNF-α receptor: IgG Fc fusion protein

INTERVENTIONS:
Drug: recombinant TNF-α receptor: IgG Fc fusion protein — 50mg weekly
  Other Names: Anbainuo

SUMMARY:
TNF- α receptor inhibitors have been used widely in practice and are well developed in China. Anbainuo is a bio-similar recombinant TNF-α receptor: IgG Fc fusion protein, approved in 2015. Up to now, Anbainuo is well applied in patients with rheumatoid arthritis (RA) or ankylosing spondylitis (AS). Although the phase II and III clinical trials both indicated that Anbainuo can effectively control the disease activity with good tolerance and safety in RA and AS patients, there is no sufficient clinical evidence in the real world. Thus, the objective of this study is to evaluate, under the actual conditions of use, dosing patterns of Anbainuo. Investigators plan to recruit 1000 adult patients with RA or AS and to follow them for 48 weeks. It is hypothesized that this study would reflect real clinical conditions (efficacy and safety assessment) of using Anbainuo in RA and AS patients.

ELIGIBILITY:
Inclusion Criteria:

* meet the diagnostic criteria of the American College of Rheumatology (ACR) (1987);
* or meet the diagnostic criteria of ankylosing spondylitis (New York, modified in 1984);
* older than 18;
* Prepare to or already start to use Anbainuo.

Exclusion Criteria:

* any acute or chronic infection or the history of active tuberculosis
* pregnant women or breast feeding women;
* malignant tumor;
* moderate to severe congestive heart failure (New York Heart Association, 3-4 grade);
* allergic to Anbainuo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA and AS patients from 30 centers (hospital) in China.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-08-24 (Estimated); Primary Completion 2020-07-24 (Estimated); Study Completion 2020-12-24 (Estimated)

PRIMARY OUTCOMES:
Percent of participants achieving clinical remission defined as a DAS28 ≥1.2 | Up to week 48
  The DAS28 is a combined index for measuring disease activity in rheumatoid arthritis (RA). The index includes swollen joint counts (SJC) and tender joint counts (TJC), both scored 0-28 (higher scores indicate higher disease activity), as well as acute phase response (APR) determined as erythrocyte sedimentation rate (ESR), and general health (GH), both scored 1-100 (higher scores indicate higher disease activity). DAS28 was calculated according to the following formula: DAS28 equals (=) [0.56 multiplied by (*) the square root (√) of TJC] plus (+) [0.28 * √ of SJC] + (0.70 * the natural logarithm (ln) ESR in millimeters per hour (mm/h)] + [0.014 * GH in mm visual analogue assessment (VAS)]. A negative change from randomization indicated improvement.
Percent of participants achieving bath ankylosing spondylitis disease activity index (BASDAI) 50 response. | Up to week 48
  BASDAI subject assessment of discomfort, pain and fatigue was measured using a 100 millimeter Visual Analog Scale (VAS); range: 0=none to 100=very severe. BASDAI 50 response defined as at least a 50 percent (%) improvement (decrease) from baseline to observation (last observation carried forward) in the BASDAI. Baseline score minus score at observation divided by Baseline score * 100 = >=50%.

SECONDARY OUTCOMES:
Change From baseline in the modified total Sharp score to week 48 | baseline and week 48
  he modified total sharp score is the sum of the erosion score (ES) and the joint space narrowing (JSN) score and has a range of 0 to 398. The ES is the sum of joint scores collected for 46 joints and has a range of 0 to 230. The JSN is the sum of joint scores collected for 42 joints and has a range of 0 to 168. A score of 0 would indicate no change and higher scores represent a worsening of joint erosions and joint space narrowing.